CLINICAL TRIAL: NCT01921179
Title: Rehabilitation of Executive Functioning in Veterans With PTSD and Mild TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: D1111-I
Record Dates: First submitted 2013-08-02; First posted 2013-08-13 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Post Traumatic Stress Disorder; Mild Traumatic Brain Injury, Concussion
Keywords: Post Traumatic Stress Disorder,; Mild Traumatic Brain Injury; Concussion; Cognitive Rehabilitation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Concussion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GOALS (Goal-Oriented Attentional Regulation) (Experimental): Goal-Oriented Attentional Regulation (GOALS) will involve 5-weeks of training (20 hours of group training (2 hour sessions, 2 days per week), 3 hours of individual training (1 hour at the beginning, halfway through and at the end of training), and approximately 20 hours of home practice). Some subjects will only receive the GOALS intervention.
  Interventions: Behavioral: GOALS (Goal-Oriented Attentional Regulation)
- EDU (Brain Health Education) (Active Comparator): Brain Health Education (EDU) will involve 5-weeks of training (20 hours of group training (2 hour sessions, 2 days per week), 3 hours of individual training (1 hour at the beginning, halfway through and at the end of training), and approximately 20 hours of homework). The EDU intervention involves education on brain health and functioning in a classroom format, with study materials for homework. Some subjects will start with EDU and then cross-over to the GOALS.
  Interventions: Behavioral: EDU (Brain Health Education)

INTERVENTIONS:
Behavioral: GOALS (Goal-Oriented Attentional Regulation) — Goal-Oriented Attentional Regulation (GOALS) will involve 5-weeks of training (20 hours of group training (2 hour sessions, 2 days per week), 3 hours of individual training (1 hour at the beginning, halfway through and at the end of training), and approximately 20 hours of home practice). Some subjects will only receive the GOALS intervention.
  Arms: GOALS (Goal-Oriented Attentional Regulation)
Behavioral: EDU (Brain Health Education) — Brain Health Education (EDU) will involve 5-weeks of training (20 hours of group training (2 hour sessions, 2 days per week), 3 hours of individual training (1 hour at the beginning, halfway through and at the end of training), and approximately 20 hours of homework). The EDU intervention involves education on brain health and functioning in a classroom format, with study materials for homework. Some subjects will start with EDU and then cross-over to the GOALS.
  Other Names: EDU
  Arms: EDU (Brain Health Education)

SUMMARY:
One of the most pressing concerns within the VA currently is the provision of interventions that address the cognitive as well as emotional problems faced by Veterans with concurrent mild TBI and PTSD. One purpose of this study is to learn more about how PTSD and mild brain injury influences how people think, act, and feel. This may include how people pay attention, keep information in memory, organize plans for achieving important goals, and manage stress. Another purpose of this research is to learn more about the effects of cognitive training on the thinking, behavior, and emotions of individuals with PTSD and mild brain injury - both in the short- and long-term. With this research, the investigators hope to better understand and treat cognitive and emotional difficulties that can occur due to PTSD and mild brain injury.

DETAILED DESCRIPTION:
The overall aim of this proposal is to investigate the potential short and long term effectiveness of a cognitive training program Goal-Oriented Attentional Self-regulation (GOALS) that targets executive control functions in Veterans with co-morbid posttraumatic stress disorder (PTSD), history of mild traumatic brain injury (mTBI), and cognitive difficulties. Both PTSD and a history of mild TBI are prevalent in Veterans from the Operation Enduring Freedom (OEF) and Operation Iraqi Freedom (OIF) conflicts, with reported rates for each disorder ranging from 14 - 22%. Both PTSD and TBI have been associated with cognitive dysfunction which may lead to functional impairment and poor community reintegration. PTSD can be highly debilitating not only due to emotional dysregulation, but also due to deficits in the cognitive control processes.

Goal-Oriented Attentional Self-Regulation (GOALS) is a therapist administered cognitive rehabilitation training that targets executive control functions of applied mindfulness-based attention regulation and goal management, and links them to participant-defined real-life goals. In a prior study with individuals with chronic brain injury, this training has improved cognitive performance in areas of complex attention / executive function, memory, complex functional task performance, and daily functioning. Furthermore, functional MRI results after training indicated significantly enhanced modulation of neural processing in extrastriate cortex and changes in prefrontal cortex. Preliminary results from a recently completed study with Veterans with a history of chronic TBI also support improvements post GOALS on neuropsychological measures of attention and executive function, performance on complex 'real-life' tasks, and self-report measures of functional performance. Furthermore, participants also showed improvement on the emotional regulation self-report measures. These findings suggest that improving cognitive control may also improve functioning in other domains such as emotional regulation and functional performance in daily life.

In a randomized, controlled intervention study design, 42 Veterans with a diagnosis of PTSD, history of mTBI and residual cognitive difficulties will participate in experimental (GOALS), and/or active comparison (Brain Health Education - EDU) interventions matched for time and intensity. Participants will be randomized to start with either 5 weeks of GOALS or EDU training. Those who begin with EDU will cross-over to GOALS, while those begin with GOALS will have 5 weeks of self-driven practice only. Both groups will participate in pre and post intervention measurements at baseline, weeks 5 and 10. Long-term follow-up will be at 6 months. Pre- and post-intervention measurements will include performance on untrained: neuro-cognitive tests assessing targeted and non-targeted cognitive domains, complex functional task performance in low structure 'real-world' setting, and self-report measures of emotional regulation and daily functioning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD
* History of mild TBI, including concussion > 6 months ago
* Cognitive difficulties affecting daily functioning
* Age 18-75
* Veteran
* At least 12th grade education or equivalent

Exclusion Criteria:

* Amnesic/Severe memory problems
* Active Substance Abuse/Dependence
* Medical condition that may affect mental status/disrupt study participation
* Active psychotropic medication changes
* Participation in evidence-based PTSD treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-07-31 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Novakovic-Agopian, PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (2):
- United States (2):
  - Martinez Outpatient Clinic and Community Living Center, Martinez, CA, Martinez, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
Following study completion and publication of results we will explore available mechanisms for data sharing

REFERENCES:
- [Result] Novakovic-Agopian T, Chen AJ, Rome S, Abrams G, Castelli H, Rossi A, McKim R, Hills N, D'Esposito M. Rehabilitation of executive functioning with training in attention regulation applied to individually defined goals: a pilot study bridging theory, assessment, and treatment. J Head Trauma Rehabil. 2011 Sep-Oct;26(5):325-38. doi: 10.1097/HTR.0b013e3181f1ead2. PMID 21169860
- [Result] Chen AJ, Novakovic-Agopian T, Nycum TJ, Song S, Turner GR, Hills NK, Rome S, Abrams GM, D'Esposito M. Training of goal-directed attention regulation enhances control over neural processing for individuals with brain injury. Brain. 2011 May;134(Pt 5):1541-54. doi: 10.1093/brain/awr067. Epub 2011 Apr 22. PMID 21515904
- [Result] Novakovic-Agopian T, Chen AJ, Rome S, Rossi A, Abrams G, D'Esposito M, Turner G, McKim R, Muir J, Hills N, Kennedy C, Garfinkle J, Murphy M, Binder D, Castelli H. Assessment of subcomponents of executive functioning in ecologically valid settings: the goal processing scale. J Head Trauma Rehabil. 2014 Mar-Apr;29(2):136-46. doi: 10.1097/HTR.0b013e3182691b15. PMID 23076096
- [Result] Novakovic-Agopian T, Kornblith E, Abrams G, Burciaga-Rosales J, Loya F, D'Esposito M, Chen AJW. Training in Goal-Oriented Attention Self-Regulation Improves Executive Functioning in Veterans with Chronic Traumatic Brain Injury. J Neurotrauma. 2018 Dec 1;35(23):2784-2795. doi: 10.1089/neu.2017.5529. Epub 2018 Jul 23. PMID 29717652

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 76 enrolled participants: 12 were excluded after in person screening for not meeting inclusion criteria CAPS diagnosis of PTSD (n=11), or substance abuse (n=1); 8 participants left study after consent for scheduling, medical/family issues; and 10 left study during baseline assessment (were not randomized)
  46 participants were randomized
Groups:
- GOALS (Goal-Oriented Attentional Regulation): Goal-Oriented Attentional Regulation (GOALS) executive training involved 5-weeks of training (20 hours of group training (2 hour sessions, 2 days per week), 3 hours of individual training, and approximately 20 hours of home practice. Participants randomized to the GOALS intervention, did no receive EDU training.
Period: 5 Week Randomized GOALS vs EDU Training
Arm/Group | GOALS (Goal-Oriented Attentional Regulation) | EDU (Brain Health Education)
Started | 24 | 22
Completed | 21 | 19
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3
Period: Long Term Follow-up After GOALS Training
Arm/Group | GOALS (Goal-Oriented Attentional Regulation) | EDU (Brain Health Education)
Started | 34 | 0 (13 out of 19 participants who completed EDU, also completed GOALS training)
Completed | 32 | 0
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- GOALS (Goal-Oriented Attentional Regulation): Goal-Oriented Attentional Regulation (GOALS) executive training involved 5-weeks of training (20 hours of group training (2 hour sessions, 2 days per week), 3 hours of individual training, and approximately 20 hours of home practice.
  Participants randomized to GOALS intervention, did no receive EDU training after completion of GOALS.
- EDU (Brain Health Education): Brain Health Education (EDU) involved 5-weeks of training (20 hours of group training , 3 hours of individual training ,and approximately 20 hours of homework). The EDU intervention involves education on brain health and functioning in a classroom format, with study materials for homework.
  Some subjects who completed EDU training during the randomized phase, completed additional 5 weeks of GOALS training.
- Total: Total of all reporting groups
Arm/Group | GOALS (Goal-Oriented Attentional Regulation) | EDU (Brain Health Education) | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (13.95) | 47.53 (14.86) | 45.08 (14.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 20 | 15 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 2
  Native Hawaiian or Pacific Islander | 1 | 1 | 2
  Black | 2 | 2 | 4
  White | 14 | 14 | 28
  More than one race | 2 | 1 | 3
  Hispanic or Latino | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 19 | 40
Attention/Executive Function Overall Z Score [Mean (Standard Deviation); unit: z score] — Attention and Executive Function Overall Domain Z Score is calculated as the average of z scores of following tests: Letter Number Sequencing, Auditory Consonant Trigrams, Digit Vigilance, Trails B, DKEFS Stroop Inhibition, DKEFS Stroop Inhibition-Switching, DKEFS Verbal Fluency Switching, DKEFS Visual Fluency Switching.
  (The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the population mean. Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population)
  z score | -0.39 (0.72) | -0.38 (0.77) | -0.39 (0.72)
Goal Processing Scale (GPS) Overall Performance Score [Mean (Standard Deviation); unit: score on a scale] — Goal Processing Scale Overall Performance score (Primary functional performance outcome ) is calculated as the average of the 8 sub-domain scores including: Planning, Initiation, Maintenance of Attention, Self-Monitoring, Sequencing and Switching Attention, Flexible Problem Solving, Memory, and Execution. Minimum value is 0, maximum value is 10. Higher scores indicate better outcome.
  score on a scale | 7.17 (1.48) | 7.31 (1.44) | 7.27 (1.39)
Profile of Mood States (POMS)-Total Mood Disturbance Score [Mean (Standard Deviation); unit: z score] — Overall psychological distress will be assessed with Profile of Mood States (POMS) questionnaire Total Mood Disturbance Z Score (primary emotional regulation outcome measure).
  (The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the population mean. Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population)
  z score | -1.69 (1.57) | -1.94 (1.06) | -1.81 (1.34)

OUTCOME MEASURES:

1. Primary Outcome: Change in Performance on Neurocognitive Measure of Attention and Executive Function Post GOALS Intervention vs EDU Control Training
Description: Attention and Executive Function Overall Domain Z Score (primary neuropsychological outcome measure) is calculated as the average of z scores of following tests: Letter Number Sequencing, Auditory Consonant Trigrams, Digit Vigilance, Trails B, DKEFS Stroop Inhibition, DKEFS Stroop Inhibition-Switching, DKEFS Verbal Fluency Switching, DKEFS Visual Fluency Switching.
  (The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the population mean. Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population)
Time Frame: baseline, 5 weeks
Population: Out of 21 participants who completed GOALS, 3 participants did not complete one or more neuropsychological tests
Measure: Mean (Standard Deviation); unit: z score
Groups:
- GOALS (Goal-Oriented Attentional Regulation): Goal-Oriented Attentional Regulation (GOALS) executive training involved 5-weeks of training (20 hours of group training, 3 hours of individual training, and approximately 20 hours of home practice. GOALS is therapist administered cognitive rehabilitation training that targets executive control functions of applied mindfulness-based attention regulation and problem solving applied to participant-defined real-life goals.
  Participants randomized to the GOALS intervention, did no receive EDU training after completion of GOALS.
- EDU (Brain Health Education): Brain Health Education (EDU) involved 5-weeks of training (20 hours of group training), 3 hours of individual training, and approximately 20 hours of homework). The EDU intervention is therapist administered, and involves education on brain health and functioning in a classroom format, with study materials for homework.
  Participants randomized to EDU intervention were offered to participate in GOALS training after completion of EDU training.
Arm/Group | GOALS (Goal-Oriented Attentional Regulation) | EDU (Brain Health Education)
Number analyzed (Participants) | 18 | 19
z score | -0.03 (0.68) | -0.39 (0.72)
Statistical Analysis 1: Comparison: GOALS (Goal-Oriented Attentional Regulation) vs EDU (Brain Health Education); Test type: Equivalence — A repeated measures MANOVA was used to compare the impact of GOALS training versus the BHE training on neurocognitive performance Attention and Executive Function Overall Domain Z Score; p < 0.01, ANOVA

2. Primary Outcome: Long Term Follow-up After GOALS Training - Change in Performance on Neurocognitive Measures of Attention and Executive Function 6+ Months Post GOALS Intervention Relative to Baseline
Description: as for outcome 1
Time Frame: baseline, 6+ months after GOALS training
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | GOALS (Goal-Oriented Attentional Regulation)
Number analyzed (Participants) | 27
z score | -0.2 (0.78)
Statistical Analysis 1: Comparison: GOALS (Goal-Oriented Attentional Regulation); Test type: Equivalence — A repeated measure multivariate analysis of variance (MANOVA) was used to compare neurocognitive performance on Overall Attention /Executive Function overall score at baseline and at 6+ month post-GOALS training follow-up; p < 0.001, ANOVA; Repeated measure MANOVA was used to compare performance on neurocognitive domain scores at baseline and at 6+ month follow-up post-GOALS training

3. Secondary Outcome: Change in Performance on Complex Functional Task -Goal Processing Scale Post GOALS Intervention vs EDU Control Training
Description: Goal Processing Scale Overall Performance score (Primary functional performance outcome ) is calculated as the average of the 8 sub-domain scores including: Planning, Initiation, Maintenance of Attention, Self-Monitoring, Sequencing and Switching Attention, Flexible Problem Solving, Memory, and Execution. Minimum value is 0, maximum value is 10. Higher scores indicate better outcome.
Time Frame: baseline; 5 weeks
Population: Out of 21 participants who completed GOALS training 3 participants did not complete one or more sub-tests of GPS.
  Out of 19 participants who completed EDU training 2 participants did not complete one or more sub-tests of GPS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GOALS (Goal-Oriented Attentional Regulation) | EDU (Brain Health Education)
Number analyzed (Participants) | 18 | 17
score on a scale | 8.10 (1.10) | 7.60 (1.04)
Statistical Analysis 1: Comparison: GOALS (Goal-Oriented Attentional Regulation) vs EDU (Brain Health Education); Test type: Equivalence — A repeated measures MANOVA was used to compare the impact of GOALS training versus the BHE training on functional performance; p > 0.05, ANOVA; A repeated measures MANOVA was used to compare the impact of GOALS training versus the BHE training on functional performance

4. Secondary Outcome: Long Term Follow-up After GOALS Training - Change in Performance on Complex Functional Task -Goal Processing Scale 6+ Months Post GOALS Intervention Relative to Baseline
Description: as for outcome 3
Time Frame: baseline, 6 months post GOALS training
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GOALS (Goal-Oriented Attentional Regulation)
Number analyzed (Participants) | 24
score on a scale | 8.23 (1.20)
Statistical Analysis 1: Comparison: GOALS (Goal-Oriented Attentional Regulation); Test type: Equivalence — A repeated measure multivariate analysis of variance (MANOVA) was used to compare performance on Goal Processing Scale Overall domain scores at baseline and 6+ month post-GOALS training follow-up; p < 0.001, ANOVA

5. Secondary Outcome: Change on Self Report Measures of Emotional Regulation GOALS Post Intervention vs EDU Control Training
Description: Overall psychological distress will be assessed with Profile of Mood States (POMS) questionnaire Total Mood Disturbance Z Score (primary emotional regulation outcome measure).
  (The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the population mean. Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population)
Time Frame: baseline, 5 weeks
Population: Out of 21 participants who completed GOALS training 3 participants did not complete one or more questions on POMS Out of 19 participants who completed EDU training 2 participants did not complete one or more questions on POMS
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | GOALS (Goal-Oriented Attentional Regulation) | EDU (Brain Health Education)
Number analyzed (Participants) | 18 | 17
z score | -1.37 (1.82) | -2.09 (0.94)
Statistical Analysis 1: Comparison: GOALS (Goal-Oriented Attentional Regulation) vs EDU (Brain Health Education); Test type: Equivalence — A repeated measures MANOVA was used to compare the impact of GOALS training versus the BHE training on emotional regulation measures - POMS Total score; p < 0.05, ANOVA; A repeated measures MANOVA was used to compare the impact of GOALS versus the BHE training on emotional regulation measures - POMS Total score

6. Secondary Outcome: Long Term Follow-up Change on Self Report Measures of Emotional Regulation 6+ Months Post GOALS Intervention
Description: Overall psychological distress is assessed with Profile of Mood States (POMS) questionnaire Total Mood Disturbance Z Score (primary emotional regulation outcome measure)
  (The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the population mean. Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population)
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | GOALS (Goal-Oriented Attentional Regulation)
Number analyzed (Participants) | 25
z score | -1.01 (1.40)
Statistical Analysis 1: Comparison: GOALS (Goal-Oriented Attentional Regulation); Test type: Equivalence — A repeated measure multivariate analysis of variance (MANOVA) was used to compare participants' self-report on POMS Total Mood Disturbance overall score at baseline and 6+ month post-GOALS training follow-up; p < 0.01, ANOVA

ADVERSE EVENTS:
Time Frame: baseline to 6 month follow-up
Description: Potential risks were minimal. The research procedures involved presented no physical risk and minimal psychological risk to the subjects. The primary risk was the potential for anxiety or boredom associated with completing behavioral assessments and training interventions.
Groups:
- EDU (Brain Health Education): Brain Health Education (EDU) involved 5-weeks of training (20 hours of group training , 3 hours of individual training ,and approximately 20 hours of homework). The EDU intervention involves education on brain health and functioning in a classroom format, with study materials for homework.
  Some subjects who completed EDU training during the randomized phase, completed the additional 5 weeks of GOALS.
Arm/Group | GOALS (Goal-Oriented Attentional Regulation) | EDU (Brain Health Education)
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/22
Other Adverse Events (participants affected / at risk) | 0/37 | 0/22

LIMITATIONS AND CAVEATS:
One important limitation of this study is a relatively small sample size, which may have also resulted in our interaction analyses being under powered, possibly leading to failure to detect true effects of group on outcomes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Full Protocol (2014-11-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT01921179/Prot_SAP_000.pdf
  • Informed Consent Form (2014-11-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT01921179/ICF_001.pdf
  • Study Protocol: Study Protocol Summary Abstract (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT01921179/Prot_002.pdf